CLINICAL TRIAL: NCT01360931
Title: The Roles of Neutrophil Elastase in Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Lam Chi Leung David, University of Hong Kong
Other Study IDs: HKU_UW_11_085
Record Dates: First submitted 2011-05-19; First posted 2011-05-26 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Lung Cancer; Chronic Obstructive Pulmonary Diseases
Keywords: Lung cancer; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Small bronchial biopsy alongside with the corresponding Bronchoalveolar lavage and bronchial aspirate will be collected in the same one bronchoscopy session
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer group: Subject with histological confirmation of lung cancer
- Control group: Subjects with no diagnosis of lung cancer

SUMMARY:
Lung cancer is the leading cause of cancer death in Hong Kong. Lung adenocarcinomas is the most common type, accounting for 70% of lung cancer and the molecular target of epidermal growth factor receptor (EGFR) gene mutation at exons 18 - 21 is present in about 50% of lung adenocarcinomas. The v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (K-ras) mutations are commonly present in the other 50% that are EGFR wildtype. EGFR and K-ras mutations are found to be mutually exclusive in the same tumor. EGFR-tyrosine kinase inhibitor (TKI) can be used as treatment for EGFR mutated tumors while no specific targeted therapy can be recommended for EGFR wildtype tumors and these patients often receive chemoirradiation, which is toxic and clinical response is suboptimal. There is a need to find alternative molecular pathways/targets in EGFR wildtype lung adenocarcinomas.

Even with EGFR mutations, good clinical response to EGFR-TKI is achieved in about 70% of these patients. This would mean suboptimal targeting of the EGFR gene or the presence of alternative pathways mediating tumor progression and susceptibility to therapy. Exploration of molecular pathways in lung cancer may allow for discovery of new molecular targets for therapeutic development.

Neutrophil infiltration is frequently observed in lung cancer. Recognized similarities between neutrophils and cancer cells include (i) ability to circulate as single cells; (ii) target attachment via vascular system; (iii) target invasion. The major difference is that migrated neutrophils will undergo apoptosis while cancer cells can escape apoptosis.

This led to the postulation that neutrophils and cancer cells may share similar inflammatory cascades by secreting a similar panel of proteases, and one of these could be neutrophil elastase (NE). Animal studies demonstrated that NE from neutrophils moves into lung tumor cells and mediates lung tumor growth via degradation of Insulin receptor substrate-1 (IRS-1), leading to activation of intracellular phosphoinositide-3-kinase (PI3k) and the v-akt murine thymoma viral oncogene homolog 1 (Akt) signaling pathways and the intracellular tyrosine kinase of the platelet-derived growth factor receptor (PDGFR).

The aims of this study are to demonstrate NE activities and the subsequent signaling cascades activated in lung cancer cells, and to verify NE and its related pathway activation in clinical lung cancer specimen.

This study will conclude the roles of NE and the therapeutic potential of NE/IRS-1/PI3K/PDGFR pathways in EGFR wildtype lung adenocarinomas.

DETAILED DESCRIPTION:
Objectives

1. To demonstrate the presence of NE in vitro and the entrance into lung adenocarcinoma cells
2. To identify the intracellular mechanisms through which NE mediates its tumor proliferating effects
3. To verify the activation of NE and its related pathway component in clinical lung adenocarcinoma specimens

Background of research

Lung Cancer in Hong Kong Lung cancer is the leading cause of cancer death in Hong Kong [1]. Surgical resection for early stage lung cancer is the only curative option and advanced stage lung cancer is treated with chemoirradiation or molecular targeted agents, one of which is Epidermal Growth Factor Receptor - Tyrosine Kinase Inhibitor (EGFR-TKI). Recent advances in molecular biology of lung cancer allowed for development of these targeted therapy. However, treatment response depends on the presence of activating EGFR gene mutation, and the median response period is usually maintained for nine to twelve months, after which the tumor usually become non-responsive or resistant to EGFR-TKI.

EGFR mutation vs EGFR wildtype lung adenocarcinomas

In Asian populations including Hong Kong, EGFR mutations at exons 18 - 21 are present in up to 50% of lung adenocarcinomas, while the other 50% are EGFR wild type lung adenocarcinomas and are usually bearing K-ras gene mutations [2]. Even with the presence of activating EGFR gene mutations at exons 18 - 21, clinical response was observed in only 70% of patients with tumors bearing EGFR mutations [3]. It is apparent that in a cohort of lung adenocarcinomas, there can be the following groupings according to their EGFR gene mutation status:

(i) EGFR mutated lung adenocarcinomas (~50%)

1. with response to TKI treatment (~35%)
2. but unresponsive to TKI treatment (~15%) (ii) EGFR wildtype lung adenocarcinomas (~50%) The presence of group (i)(b) tumors with EGFR but failed response to treatment would mean suboptimal targeting of EGFR and the presence of group (ii) EGFR wildtype tumors would imply alternative pathways mediating tumor progression and susceptibility to tumor therapy in lung cancer. Exploration of molecular pathways in lung adenocarcinomas may allow for discovery of new molecular targets for therapeutic development in lung cancer.

Neutrophils vs cancer cells

Neutrophil infiltration, and hence inflammatory infiltrate, is a frequently observed in lung cancer [4]. Recognized similarities between neutrophils and cancer cells include:

1. ability to circulate as single cells
2. target attachment via vascular system
3. target invasion Neutrophils achieve migration through pulmonary epithelial layers by secreting NE, which is readily balanced by the local action of secretory leukocyte peptidase inhibitor (SLPI). SLPI has also been detected in cancer tissues but the relevant function role in lung cancer has not been defined yet [5]. The major difference between neutrophils and cancer cells lies in the fact that migrated neutrophils will undergo apoptosis while cancer cells can escape apoptosis and are able to proliferate in target organs.

The possible roles of NE in lung cancer This has led to the speculation that neutrophils and cancer cells may share similar inflammatory cascades by secreting a similar panel of proteases, and one of these had been demonstrated to be neutrophil elastase (NE). The action of NE may happen at different cellular levels: (1) action on extracellular matrix to facilitate migration and tissue invasion; (2) action on cell surface signaling receptors; or (3) intracellular action on signaling pathways following uptake into signaling endosomes. There are recent evidence in animal studies that NE secreted by neutrophils actually moved into lung tumor cells and mediates lung tumor growth via degradation of Insulin receptor substrate-1 (IRS-1) and subsequent effects on the intracellular PI3K signaling pathways acting on the intracellular tyrosine kinase domain of the platelet-derived growth factor receptor (PDGFR)[6]. It is possible that neutrophils infiltrating lung tumor stromal tissues may be acting in collaboration with cancer cells via the direct and indirect actions of NE.

Work done by others Immunoreactive NE, both in free and in complex forms, can be demonstrated in breast cancer cell lines [7] and lung cancer cell lines [8]. NE activities has been further demonstrated in human breast cancer tissues [9] but not in human lung cancer tissues or normal lung tissues. These showed that NE is present at the tissue level but their intracellular action, whether enzymatically active or signaling active, has not been delineated clearly yet.

In breast cancer tissues, the higher the amount of extracted tissue NE, the worse was the prognosis [9] and similar prognostic significance was suggested for NE in non-small cell lung cancer [10].

When lung cancer cells were inoculated into severe combined immunodeficiency (SCID) mice, concomitant administration of NE inhibitor, ONO-5046, will completely suppressed tumor growth and appearance of metastatic foci [11]. The exact mechanism of action of ONO-5046 remains to be clarified.

NE has also been shown to cleave cell surface epidermal growth factor (EGF) and transforming growth factor-alpha (TGF-α) [12, 13]. This may send aberrant signals to tumor cells EGF receptors and promote cancer cell proliferation in vitro.

TGF-α also induced NE expression in human cancer cell lines (breast and pancreas)

There were recent works by Houghton et al [6] demonstrating NE could influence lung cancer growth and development by:

1. permeating into lung tumor cells (A549 lung adenocarcinoma cell line with Kras mutation) and, via degradation of IRS-1, mediating tumor cell progression.
2. being blocked by specific inhibitors (ONO-5046), leading to aberrant intracellular signaling and then tumor cell growth arrest.

Work done by our groups NE in airway inflammation Our group had done work related to the roles of NE in airway inflammation and diseases and we have raised cancer and normal bronchial bronchial epithelial cell lines from local patients that would be appropriate models for testing the hypothesis in local patient populations.

Syndecan-1 was found to be able to bind NE in sputum sol of bronchiectasis, supporting the role of NE complexed with syndecan-1 in balance with antielastase [14]. We have also demonstrated shed syndecan-1 from human lymphoid cell line was able to bind to NE, disturbing the NE and anti-elastase balance in the airway environment, and thus could be playing a role in airway inflammation [15].

We have tried to unopposed NE in the airway fluids in a cigarette smoke-induced model of COPD in rats. Sulfated maltoheptaose to chelate NE was administered to rats and bronchoalveolar lavage fluid (BALF) and lung tissues were collected 3 days after administration that showed significant declines in NE activity and myeloperoxidase activity as compared to BALF of smoking rats not treated. Significant reduction in neutrophil accumulation was also observed in BALF and lung tissue sections. Airspace enlargement was significantly reduced following the treatment. All these results suggested that sulfated maltohepatose is a potential therapeutic against neutrophilic inflammation in the airways of patients with COPD. (unpublished data).

We have also tested the NE activity of a lung adenocarcinoma cell line A549 and found that radio-labelled cells migrate into lung cancer cells and is enzymatically inactive (unpublished data) Lung cancer cell lines and normal bronchial epithelial cells and clinical lung cancer tissue bank

We have recently established primary lung cancer and normal bronchial epithelial cell lines from local Chinese patients and they were characterized with in vitro growth kinetics, morphological and immunohistochemical studies and gene expression profiling [16]. At the moment, we have:

1. Four primary lung adenocarcinoma cell lines (HKULC 1 - 4) published [16] and six more newly established in various phase of characterization.
2. Two new normal bronchial epithelial cell lines immortalized with standard protocols with cdk4 and hTert infections [17].

These new cell lines were all derived from clinical specimen from the local Hong Kong Chinese patients and more are becoming established with continued accrual of clinical collection. The clinical data of the patients, including gender and smoking history, from which these primary lung adenocarcinoma cell lines originated were known. Together with 10 other ATCC lung adenocarcinoma cell lines and established normal bronchial epithelial lines (HBEC-KT 1 - 5) from John Minna MD, Tx, USA, these cell lines will provide invaluable materials to test for in vivo effects of NE on cancer cells.

With the collaboration of Queen Mary Hospital Cardiothoracic Surgical Department, we have also collected 40 pairs of resected lung adenocarcinomas and normal lung tissues that will allow for verification of in vitro findings in clinical specimens. Further collection accrual of clinical specimens is in progress

The research questions to be addressed (Figure 1) are:

1. What are the roles of NE in lung adenocarcinoma proliferation?
2. How are such roles of NE mediated at the intracellular signaling level? Is IRS-1/PI3K/PDGFR the most common axis involved in cancer cells? Or there will be 'cross-talk' with pathways such as EGFR or TNF-α in lung adenocarcinoma proliferation?
3. Can we verify such roles of NE in cancer proliferation in human lung adenocarcinoma tissues?

The aims of the study will be:

1. To determine the mode of entrance and site of action of labeled NE in lung adenocarcinoma cells
2. To study the activation of IRS-1/PI3K/PDGFR in lung adenocarcinoma cells after penetrance by NE and if there will be concurrent activation of other signaling pathways including the EGFR and TNF-α pathways
3. To study the effects of blocking NE with specific NE inhibitors on lung adenocarcinoma cell proliferation
4. To verify the above mechanisms of actions of NE in clinical lung adenocarcinoma specimens

Plan of study:

1. EGFR mutation profiling of lung adenocarcinoma cell lines and resected lung adenocarcinomas Genomic DNA will be extracted from available lung adenocarcinoma cell lines (20 specimens) as well as microdissected surgical lung adenocarcinoma specimens. Exons 18 - 21 will be PCR-amplified and directly sequenced to read for EGFR mutation in exons 18 - 21. This will characterize available lung adenocarcinomas cell lines and clinical tumor specimens with respect to EGFR gene mutation or EGFR wildtype for subsequent work, where experimental results will be compared between the two groups.
2. For aim (1) - (3), the mode of entrance and site of action of NE in lung adenocarcinoma cells will be studied.

   Live cell imaging Live cell imaging technique with Alex-Flour-488-labelled NE will be employed to localize and follow the path of NE entrance into lung adenocarcinoma cells. Eglin C, a proteolytic inhibitor, will be applied at the same time. Normal bronchial epithelial cell lines will be used for comparison. The intracellular location of entrance and possible activated structural changes will be recorded.

   NE-specific reverse transcription PCR cDNA amplified from total RNA will be amplified using RT-PCR with specific primers 5'-GAG GCA ATT CCG TGG ATT AG-3' and 5' ACG ACA TCG TGA TTC TCC AG-3' Western blotting NE-stimulated cells from (1) above will have proteins extracted by standard methods followed by immunoblotting with specific monoclonal antibodies to study related signaling pathways including pAkt, Akt, p85, IRS-1, IRS-2, PDGF, PDGF-α, pPDGF-α, p44/42 MAPK, phosphor-p44/42 MAPK as well as pEGFR and TNF-α. Anti-β-actin will be used as endogenous control. Reaction to individual markers will be done in triplicates Cell growth assay The effect of ONO-5046, a specific NE inhibitor, on cell growth and proliferation will be studied on lung adenocarcinoma cell lines compared to control (no drug administration).
3. For aims (4), we would like to study the activation of relevant signaling pathways upon NE stimulation

   1. Immunohistochemistry Immunohistochemical staining will be performed on clinical lung adenocarcinoma specimens with specific monoclonal antibodies against NE, PDGF, PDGFR, IRS-1 and EGFR. Concordance of staining pattern will be examined between IRS-1 and EGFR or PDGF respectively. The proportion of discordant cases will be compared with the proportion of concordant cases.
   2. NE assay in clinical lung cancer specimens from human subjects Clinical lung cancer specimens will be collected from patients with lung adenocarcinomas and NE activities assayed.

ELIGIBILITY:
Inclusion Criteria:

* All subjects undergoing clinical diagnostic or therapeutic procedures, including:

  1. Fibreoptic bronchoscopy or pleuroscopy
  2. Diagnostic or Therapeutic pleurocentesis AND who are mentally fit to give informed consent for donation of clinical specimens

Exclusion Criteria:

* Patients who cannot give written informed consent or refuse to give such consent for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing diagnostic bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The protein expression levels of biomarkers related to neutrophil elastase | Jan 2011 - June 2013 (30 months)
  The protein expression levels of phosphorylated Akt (pAkt), IRS-1, IRS-2, PDGF, mitogen activated kinase(MAPK) as well as phosphorylated EGFR (pEGFR) and TNF-α and β-actin will be assessed semi-quantitatively on electrophoretic blotting intensity.

SECONDARY OUTCOMES:
Immunohistochemical staining for NE, IRS-1 and EGFR | Jan 2011 - June 2013 (30 months)
  Fields captured from four different fields from each stained (NE, IRS-1 and EGFR) lung tumor slides will be scored as 0 = absent, 1 = weak, 2 = strong and present. In NE positive cases, concordant and discordant cases of IRS-1 vs PDGF or EGFR staining will be observed. Likelihood ratio tests determining if proportion of discordant cases was significantly larger than half the cases will be presented

CONTACTS AND LOCATIONS:
Overall Officials: David CL LAM, MBBS, FRCP(Edin), FCCP, FACP, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong